CLINICAL TRIAL: NCT02677038
Title: Olaparib for BRCAness Phenotype in Pancreatic Cancer: Phase II Study
Brief Title: Olaparib in Treating Patients With Stage IV Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0503; NCI-2016-00351 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0503 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Pancreatic Ductal Adenocarcinoma; Stage IV Pancreatic Cancer AJCC v6 and v7
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (olaparib) (Experimental): Patients receive olaparib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281

SUMMARY:
This phase II trial studies how well olaparib works in treating patients with stage IV pancreatic cancer. Olaparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of olaparib monotherapy in stage IV pancreatic ductal adenocarcinoma (PDAC) with breast cancer, early onset (BRCA)ness.

SECONDARY OBJECTIVES:

I. To further determine the efficacy of olaparib in the study population.

SAFETY OBJECTIVES:

I. To assess the safety and tolerability of olaparib.

EXPLORATORY OBJECTIVES:

I. To identify tissue based biomarkers of defective homologous recombination repair (HRD).

OUTLINE:

Patients receive olaparib orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 8 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas
* Family history: one or more close blood relative with ovarian carcinoma at any age or breast cancer age 50 or younger or two relatives with breast, pancreatic or prostate cancer (Gleason 7 or higher) at any age, or patients with Ashkenazi Jewish ancestry; however, patients with previously identified genetic aberrations that are associated with homologous recombination deficiency (HRD) will be eligible even in the absence of family history (e.g. somatic BRCA mutation, Fanconi anemia gene, ATM or RAD51 mutations)
* Patients must be germline BRCA 1 or 2 negative; (Note: if BRCA status was previously determined, that result is acceptable but documentation of status must be available; subjects with unknown status will be referred to genetic counselling for BRCA testing as per standard of care) and/or patients with previously identified genetic aberrations that are associated with HRD will be eligible even in the absence of family history (e.g. somatic BRCA mutation, Fanconi Anemia gene, ATM or RAD51 mutations)
* Patients must have received at least one prior therapy for metastatic disease to be eligible
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* All treated patients have the option to undergo pre-treatment biopsy (liver, omentum, lung or lymph node) to be eligible
* Patients with prior malignancy and treated with no evidence of active disease, and more than 2 years from initial diagnosis are eligible
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Karnofsky > 70)
* Leukocytes >= 3,000 cells/mm^3
* Absolute neutrophil count >= 1,500 cells/mm^3
* Platelets >= 75,000 cells/mm^3
* Hemoglobin >= 9 g/dl (no blood transfusions within 4 weeks prior to enrollment)
* Total bilirubin < 1.5 x institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x IULN without liver metastasis; =< 5 x IULN for patients with liver metastasis
* Creatinine not greater than upper institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* International normalized ratio (INR) < 1.5
* Women of childbearing potential (defined as not post-menopausal for 12 months or no previous surgical sterilization) and fertile men must agree to use two highly effective forms of contraception while they are receiving study treatment and for 30 days after last dose of study drug; male subjects must agree to refrain from sperm donation during the study and for 30 days after the last dose of study drugs
* Ability to understand and the willingness to sign a written informed consent document; signed informed consent form must be obtained prior to initiation of study evaluations and/or activities

Exclusion Criteria:

* Uncontrolled intercurrent illness including symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia and myocardial infarction (MI) within 3 months of initiation of therapy
* Patients whose tumors are deemed to be platinum-refractory will be excluded from the trial
* Pregnancy or lactation
* Patient has active and uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
* Patient has undergone major surgical resection within 4 weeks prior to enrollment
* Patient received radiotherapy, surgery, chemotherapy, or an investigational therapy within 2 weeks prior to study entry
* Patient has serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive an experimental research drug
* Serious psychiatric or medical conditions that could interfere with treatment
* Major bleeding in the last 4 weeks prior to study entry
* Concomitant use of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors
* Resting electrocardiogram (ECG) with corrected QT interval (QTc) > 470 msec (Fridericia's scale)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milind Javle, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 patients were recruited at MD Anderson Cancer Center Houston Tx USA
Groups:
- Olaparib Monotherapy in Advanced Previously Treated PDAC With BRCAness: Eligible patients received 300mg Olaperib tablet twice daily until investigator assessed objective radiologic disease progression, toxic effects or patient withdrawal.
Period: Overall Study
Arm/Group | Olaparib Monotherapy in Advanced Previously Treated PDAC With BRCAness
Started | 24
Completed | 22
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Olaparib Monotherapy in Advanced Previously Treated PDAC With BRCAness
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 62 [46 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The primary endpoint was the objective response rate assessed by the investigator using the modified RECIST v1.1 criteria.
Time Frame: 5 years 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib Monotherapy in Advanced Previously Treated PDAC With BRCAness
Number analyzed (Participants) | 22
Participants
  Partial Response | 1
  Stable Disease | 15

2. Secondary Outcome: Progression Free Survival
Description: The Progression Free Survival defined as the time from enrollment until radiologic disease progression and it is assessed by the investigator review using modified RECIST v1.1 criteria or by death by any cause. This was applied to all patients from MD Anderson Cancer Center Houston Tx USA.
Time Frame: 5 years 8 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib Monotherapy in Advanced Previously Treated PDAC With BRCAness
Number analyzed (Participants) | 22
Months | 4.83 [3.61 to 7.82]

3. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the time from the date of enrollment to the date of death or last follow up. This was applied to all patients from MD Anderson Cancer Center Houston Tx USA
Time Frame: 5 years 8 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib Monotherapy in Advanced Previously Treated PDAC With BRCAness
Number analyzed (Participants) | 22
Months | 16.1 [13.5 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: 5 years, 8 months
Arm/Group | Olaparib Monotherapy in Advanced Previously Treated PDAC With BRCAness
All-Cause Mortality (participants affected / at risk) | 10/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 22/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olaparib Monotherapy in Advanced Previously Treated PDAC With BRCAness (N=22)
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 13
Alanine aminotransferase increased (Investigations) | 9
Alkaline phosphatase increased (Investigations) | 13
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 19
Anorexia (Metabolism and nutrition disorders) | 12
Anxiety (Psychiatric disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Ascites (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 9
Bile duct stenosis (Hepatobiliary disorders) | 1
Biliary tract infection (Infections and infestations) | 1
Bloating (Gastrointestinal disorders) | 2
Blood bilirubin increased (Investigations) | 3
Bruising (Injury, poisoning and procedural complications) | 1
Chest pain - cardiac (Cardiac disorders) | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Chills (Gastrointestinal disorders) | 5
Colitis (Gastrointestinal disorders) | 1
Conjunctivitis (Infections and infestations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Creatinine increased (Investigations) | 4
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 11
Dizziness (Nervous system disorders) | 9
Duodenal ulcer (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Edema limbs (General disorders) | 3
Edema trunk (General disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Esophagitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 22
Fever (General disorders) | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Flu like symptoms (General disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Gastrointestinal pain (Gastrointestinal disorders) | 1
General disorders and administration site conditions - (Other), specify (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
GGT increased (Investigations) | 12
Headache (Nervous system disorders) | 3
Hematuria (Renal and urinary disorders) | 2
Hepatobiliary disorders - (Other), specify (Hepatobiliary disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 10
Hyponatremia (Metabolism and nutrition disorders) | 4
Insomnia (Psychiatric disorders) | 8
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Localized edema (General disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Nausea (Gastrointestinal disorders) | 16
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Neutrophil count decreased (Investigations) | 3
Non-cardiac chest pain (General disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Palpitations (Cardiac disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 3
Platelet count decreased (Investigations) | 7
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Presyncope (Nervous system disorders) | 1
Proteinuria (Renal and urinary disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2
Psychiatric disorders - (Other), specify (Psychiatric disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Sinus bradycardia (Cardiac disorders) | 2
Somnolence (Nervous system disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Thromboembolic event (Vascular disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Urinary frequency (Renal and urinary disorders) | 3
Urinary tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 6
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT02677038/Prot_SAP_000.pdf